CLINICAL TRIAL: NCT04962100
Title: Capacitation-associated Protein Tyrosine Phosphorylation As a Possible Biomarker of Sperm Selection in Sperm from Patients and Donors
Brief Title: Capacitation-associated Protein Tyrosine Phosphorylation As a Possible Biomarker of Sperm Selection
Acronym: FOSFOTIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1608-SEV-065-CG
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Sperm Capacitation
Keywords: Capacitation; Tyrosine phosphorylation; Flow cytometry; Biomarker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study population (Experimental): Male patients and donors who provide a sample of fresh ejaculated semen will be the population of this study, as well as female patients undergoing artificial insemination with their partner's semen or frozen donor semen.
  Interventions: Other: Analysis of capacitation-associated tyrosine phosphorylation in human sperm by flow cytometry

INTERVENTIONS:
Other: Analysis of capacitation-associated tyrosine phosphorylation in human sperm by flow cytometry — After the assessment of the macroscopic and microscopic characteristics of the sample, we will wash the sample and process it using three layers of density gradients.
  In the case of samples for diagnostic analysis, the remaining volume will be incubated in at 37ºC, and 0.1-0.2 ml aliquots will be taken from the end of the processing at t0 (just before introducing the sample in the incubator), at t1 (after one hour of incubation) and at t3 (after 3 hours of incubation). Additionally, a sample will be taken after washing, prior to processing the sample with the density gradients. In the case of samples processed for insemination, an additional aliquot will be taken at the exact moment in which the insemination is carried out and the elapsed incubation time will be noted.
  The evaluation of the capacitation will be carried out by analyzing the state of phosphorylation of tyrosines by flow cytometry.

SUMMARY:
Sperm undergo complex selection processes and physiological changes as they move through the female reproductive tract. Ejaculated-sperm must undergo a set of molecular and biochemical changes globally named as capacitation in order to acquire the ability to fertilize the oocyte. These changes include post-translational modifications of sperm proteins, with phosphorylation of tyrosine residues being one of the most outstanding characteristics of the capacitation process. In the laboratory, the capacitation process is recreated artificially before performing artificial insemination or in vitro fertilization treatments. The sample is then incubated until it is used in the treatment. Reproductive success rates can be affected by differences in incubation times and levels of capacitation of the sample. In this study, the investigators intend to study the capacitation state of the sample by measuring the levels of phosphorylation of the tyrosine residues of the proteins contained in the sperm that have already been subjected to the capacitation process in vitro.

DETAILED DESCRIPTION:
The human male deposits millions of sperm cells in the woman's vagina at the time of ejaculation. However, only a few sperm cells are able to reach the fallopian tubes. In fact, only between 100-1000 sperm will reach the cumulus-oocyte complex and only one will be able to fertilize the oocyte.

The sperm cells from the ejaculate of all mammals are unable to fertilize the oocyte. In order to acquire the fertilization competence, sperm must undergo a process called capacitation. Capacitation has been defined as a complex phenomenon that involves biochemical and physiological changes in the sperm.

These changes are such as:

* Loss of proteins or replacement by others of lower molecular weight
* Transformation of phospholipids, decreased cholesterol/phospholipid ratio
* Changes in the carbohydrate fraction of glycoproteins
* Lipid and protein mobility

Not all the events involved in the complex capacitation process are known.

The following stages can be differentiated:

* Cell membrane fluidification
* Increased intracellular Ca2+
* Generation of controlled amounts of reactive oxygen species
* Increased intracellular pH and hyperpolarization of sperm membrane potential
* Protein phosphorylation (serine, threonine and tyrosine residues)

Under in vivo conditions, motile sperm actively migrate through the cervical mucus and are separated from the rest of the ejaculate. In vitro, sperm capacitation can be achieved if they are subjected to particular culture conditions during the necessary period of time.

After capacitation, sperm acquires three characteristics:

1. Hyperactivation.
2. Acrosomic reaction.
3. Sperm-oocyte interaction.

The capacitation process is necessary for the sperm to be able to cross the layer of cells that surround the oocyte and to undergo the acrosome reaction. Only a fraction of sperm are known to reach the capacitation state at some point.

The capacitation process depends mainly on post-translational modifications of proteins. One of the most important modifications that these proteins undergo is phosphorylation. During sperm capacitation, serine, threonine and tyrosine residues are phosphorylated. However, phosphorylation of tyrosine residues is the best indicator of sperm capacitation.

The evaluation of the phosphorylation of the tyrosine residues of the sperm proteins by flow cytometry makes it possible to assess the degree of capacitation of the sperm in vitro and to determine how many of them have carried out this process adequately . As previously mentioned, not all sperm cells of a sample undergo the capacitation process and not all of them present the same percentage of phosphorylated proteins in tyrosine residues.

Certain events, such as the cryopreservation process and the incubation times of the samples until their use in fertility treatments (IA or IVF / ICSI), can affect the capacitation process. Therefore, the measurement of the levels of tyrosine phosphorylation of the sperm by flow cytometry can allow the investigators to know the level of capacitation of the sample. There are studies that report changes in success rates when samples are incubated different period of times. The incubation period affects the rate of acrosomal reaction of sperm and may even affect DNA fragmentation. Furthermore, the temperature at which such incubation is carried out also seems to affect sperm capacitation.

Based on the above, this project aims to analyze the possible correlation between the levels of tyrosine phosphorylation in sperm and the functional quality of the seminal sample, as well as the reproductive success of the cycle. In parallel, the investigators will analyze whether the sperm capacitation process is affected by the incubation times of the sample once it has been capacitated or whether it depends exclusively on the quality of the seminal sample and is intrinsic to the male.

ELIGIBILITY:
Inclusion criteria:

* To have signed the written informed consent before starting any procedure related to the study.
* Sexual abstinence (2 to 5 days).
* To be a male patient who delivers a fresh seminal sample for diagnosis or artificial insemination treatment.
* To be a male donor who delivers a fresh seminal sample for donation or for previous tests to include him in the donation programme.
* To be a female patient undergoing artificial insemination.

Exclusion criteria:

* Use of sperm of testicular or epididymal origin.
* Cryptozoospermia or oligozoospermia with sperm concentration <1 mill/ml.
* Ejaculates obtained with more than 5 days of sexual abstinence.
* Frozen semen samples for artificial insemination cycles with partner's semen.
* Female patients who present uterine malformations that compromise the viability of the pregnancy (intramural or submucosal fibroids > 3 cm, polyps, adenomyosis or congenital or acquired malformations). Female patients with hydrosalpinx.
* Patients who have suffered two or more previous abortions (repeated abortions).
* Patients with a body mass index greater than 30 Kg / m2.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
To determine the state of sperm capacitation by assessing the phosphorylation of tyrosine residues | 1 day
  Flow cytometry analysis will be carried out to evaluate the levels of phosphorylation of tyrosine residues in sperm proteins of seminal samples capacitated in vitro in order to determine their capacitation statuscytometry of seminal samples capacitated in vitro in order to determine their capacitation status

CONTACTS AND LOCATIONS:
Overall Officials: Cristina González Ravina, PhD, Principal Investigator — IVI RMA Sevilla
Locations (1):
- IVI RMA Sevilla, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available to other researchers.
Supporting Information: CSR
Time Frame: The IPD and any additional supporting information will become available after the analysis of the data and publication of the study results.
Access Criteria: Scientific article

REFERENCES:
- [Background] Said TM, Land JA. Effects of advanced selection methods on sperm quality and ART outcome: a systematic review. Hum Reprod Update. 2011 Nov-Dec;17(6):719-33. doi: 10.1093/humupd/dmr032. Epub 2011 Aug 25. PMID 21873262
- [Background] Aitken RJ, Nixon B. Sperm capacitation: a distant landscape glimpsed but unexplored. Mol Hum Reprod. 2013 Dec;19(12):785-93. doi: 10.1093/molehr/gat067. Epub 2013 Sep 26. PMID 24071444
- [Background] Bianchi E, Doe B, Goulding D, Wright GJ. Juno is the egg Izumo receptor and is essential for mammalian fertilization. Nature. 2014 Apr 24;508(7497):483-7. doi: 10.1038/nature13203. Epub 2014 Apr 16. PMID 24739963
- [Background] Henkel R. Sperm preparation: state-of-the-art--physiological aspects and application of advanced sperm preparation methods. Asian J Androl. 2012 Mar;14(2):260-9. doi: 10.1038/aja.2011.133. Epub 2011 Dec 5. PMID 22138904
- [Background] Visconti PE, Bailey JL, Moore GD, Pan D, Olds-Clarke P, Kopf GS. Capacitation of mouse spermatozoa. I. Correlation between the capacitation state and protein tyrosine phosphorylation. Development. 1995 Apr;121(4):1129-37. doi: 10.1242/dev.121.4.1129. PMID 7743926
- [Background] Visconti PE. Understanding the molecular basis of sperm capacitation through kinase design. Proc Natl Acad Sci U S A. 2009 Jan 20;106(3):667-8. doi: 10.1073/pnas.0811895106. Epub 2009 Jan 14. No abstract available. PMID 19144927
- [Background] Liu DY, Clarke GN, Baker HW. Tyrosine phosphorylation on capacitated human sperm tail detected by immunofluorescence correlates strongly with sperm-zona pellucida (ZP) binding but not with the ZP-induced acrosome reaction. Hum Reprod. 2006 Apr;21(4):1002-8. doi: 10.1093/humrep/dei435. Epub 2006 Jan 20. PMID 16428332
- [Background] Kumaresan A, Siqueira AP, Hossain MS, Johannisson A, Eriksson I, Wallgren M, Bergqvist AS. Quantification of kinetic changes in protein tyrosine phosphorylation and cytosolic Ca(2)(+) concentration in boar spermatozoa during cryopreservation. Reprod Fertil Dev. 2012;24(4):531-42. doi: 10.1071/RD11074. PMID 22541541
- [Background] Escoffier J, Navarrete F, Haddad D, Santi CM, Darszon A, Visconti PE. Flow cytometry analysis reveals that only a subpopulation of mouse sperm undergoes hyperpolarization during capacitation. Biol Reprod. 2015 May;92(5):121. doi: 10.1095/biolreprod.114.127266. Epub 2015 Apr 8. PMID 25855261
- [Background] Naresh S, Atreja SK. The protein tyrosine phosphorylation during in vitro capacitation and cryopreservation of mammalian spermatozoa. Cryobiology. 2015 Jun;70(3):211-6. doi: 10.1016/j.cryobiol.2015.03.008. Epub 2015 Mar 28. PMID 25828199
- [Background] Mansour RT, Serour MG, Abbas AM, Kamal A, Tawab NA, Aboulghar MA, Serour GI. The impact of spermatozoa preincubation time and spontaneous acrosome reaction in intracytoplasmic sperm injection: a controlled randomized study. Fertil Steril. 2008 Sep;90(3):584-91. doi: 10.1016/j.fertnstert.2006.11.176. Epub 2008 Mar 4. PMID 18295761
- [Background] Zhang XD, Chen MY, Gao Y, Han W, Liu DY, Huang GN. The effects of different sperm preparation methods and incubation time on the sperm DNA fragmentation. Hum Fertil (Camb). 2011 Sep;14(3):187-91. doi: 10.3109/14647273.2011.604817. Epub 2011 Aug 23. PMID 21859363
- [Background] Marin-Briggiler CI, Tezon JG, Miranda PV, Vazquez-Levin MH. Effect of incubating human sperm at room temperature on capacitation-related events. Fertil Steril. 2002 Feb;77(2):252-9. doi: 10.1016/s0015-0282(01)02982-x. PMID 11821080